CLINICAL TRIAL: NCT01583153
Title: Randomised Controlled Trial Comparing Hospital Inpatient vs Home Rehabilitation After Total Knee
Brief Title: The HIHO Study: Hospital Inpatient vs Home Rehabilitation After Total Knee Replacement
Acronym: HIHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mark Buhagiar (Other)
Collaborators: HammondCare (Unknown)
Responsible Party: Sponsor-Investigator, Mark Buhagiar, Manager of Allied Health, Principal Investigator, South West Sydney Local Health District
Organization: South West Sydney Local Health District (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HIHO-1042554
Record Dates: First submitted 2012-04-19; First posted 2012-04-23 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hospital Inpatient Rehabilitation (HI) (Active Comparator)
  Interventions: Other: Hospital Inpatient Rehabilitation
- Hybrid Home Programme (HO) (Active Comparator)
  Interventions: Other: Hybrid Home Programme (HO)

INTERVENTIONS:
Other: Hospital Inpatient Rehabilitation — Those allocated to HI will be admitted to the adjacent rehabilitation hospital, Braeside Rehabilitation Hospital, for 10 days. As per the private sector, HI participants will receive twice-daily supervised physiotherapy comprising 1-1.5 hr class-based exercises and 1-1.5 hr one-to-one therapy. Prior to discharge, participants will be familiarised with the home programme as described in second arm. All participants will be required to complete a diary detailing programme adherence, healthcare utilisation, and social costs relating to carer-burden. Participants will attend the group-based sessions as per HO below for monitoring and progression of programme. An additional FIM outcome measure will be taken for this arm on admission and discharge from the inpatient rehab unit.
  Arms: Hospital Inpatient Rehabilitation (HI)
Other: Hybrid Home Programme (HO) — The HO will be based on what is standard care in the local health district and guidelines for exercise in the elderly and those with osteoarthritis. Approximately 2 weeks post-surgery, participants allocated to the HO will attend 1 group-based exercise session in the Physiotherapy Department (Fairfield Hospital) where the home programme will be rehearsed and exercises individualised as required due to co-morbidities. The programme comprises general aerobic components as well as general functional and muscle-specific exercises focused on restoring knee mobility, lower limb strength, and normal neuromuscular co-ordination and gait patterns. Participants will be able to return for 2-3 sessions over the 6-week period.
  Arms: Hybrid Home Programme (HO)

SUMMARY:
Total knee replacement (TKR) surgery is a common and highly effective treatment option for alleviating the pain and disability caused by chronic arthritis. The associated rehabilitation costs, however, impose a significant burden on the health system. In particular, inpatient rehabilitation - utilised by approximately 43% of private TKR recipients in NSW and 29% Australia-wide is of greatest concern, costing, on average, $7000 (AU) per inpatient episode.

The overarching aim of this study is to establish whether inpatient rehabilitation is necessary after TKR for patients with osteoarthritis (OA) who could otherwise be discharged directly home.

The main hypothesis to be tested by the proposed study is that TKR recipients who receive inpatient rehabilitation in addition to participating in a home programme, compared to patients who participate in a home programme only, will achieve a superior level of mobility. If superiority is shown, a cost-effectiveness analysis will be undertaken.

Secondary hypotheses to be tested relate to patient-reported knee pain and function, health-related quality of life, functional ambulation, and knee joint mobility.

Superiority in these outcomes will be evident at six months after surgery.

DETAILED DESCRIPTION:
As preferences for therapy can be a confounder in RCTs, patients will be asked their preference for rehabilitation post TKR, prior to randomisation.

Patients will be randomised once a hospital bed is available.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients presenting for elective, primary, unilateral TKR at the Whitlam Joint Replacement Centre (Fairfield Hospital) will be screened for eligibility at the pre-admission clinic by the study Project Manager (PM).
* primary diagnosis of OA

Exclusion Criteria:

* predisposition for requiring prolonged inpatient supervision (eg requiring assistance with at least one personal activity of daily living or lack of social support)
* inability to comprehend the study protocol.
* catastrophic complication arising post-surgery which precludes rehabilitation commencing within 2-3 weeks of surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2012-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Walking distance at 6 months post surgery, measured using the Six-Minute Walk Test (6MWT) | Pre surgery; 10 weeks, six months and twelve months after surgery.
  Functional mobility is a composite of several factors targeted in rehabilitation programs after TKA such as lower limb strength, knee range of motion, and balance. Second, a functional outcome is more likely to be directly influenced by the intervention (rehabilitation), and the intervention aims to improve walking. Third, the 6MWT is highly reproducible within the individual. Fourth, it is likely to be less susceptible to misinterpretation and less culturally sensitive than patient-reported outcomes. Fifth, the test does not appear to suffer from the floor or ceiling effects associated with many patient-reported outcomes. Sixth, an observer-measured outcome is less likely to be influenced by a preference effect compared to a patient-reported outcome, and this is particularly important when the intervention under examination cannot be blinded from the recipient. Together, these attributes mean the results for our primary outcome should be readily translatable to any TKA cohort.

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Pre surgery; 10 weeks, six months and twelve months after surgery.
Knee range of motion | Pre surgery; 10 weeks, six months and twelve months after surgery.
EQ5D | Pre surgery; 10 weeks, six months and twelve months after surgery.
  The EQ5D is a standardised measure providing a simple, generic measure of health. It looks at mobility, self-care, usual activities, pain/discomfort and anxiety/depression, and provides a simple descriptive profile and a single index value for health status.
Cost of surgery | Pre surgery; 10 weeks, six months and twelve months after surgery.
  Itemised list of health service use, expenditure and days off work
Patient preference for therapy | After consenting to participation and prior to randomisation
  Typical demographic and complication data (such as re-admission, re-operation, knee manipulation, death, venous thrombo-embolism, wound infection) will also be collected. As preferences for therapy can be a confounder in RCTs, patients will be asked their preference for rehabilitation post TKR prior to randomisation. Question may be 'What is your preference for rehab? Is it home based, inpatient or no preference?
15 metre walk test | Pre surgery; 10 weeks, six months and twelve months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Justine M Naylor, PhD BAppSc(Phty), Principal Investigator — SWSLHD; Ian A Harris, PhD, MBBS, M Epi, Principal Investigator — SWSLHD; Friedbert Kohler, Principal Investigator — HammondCare; Mark Buhagiar, MHM BAppSc(Phty), Principal Investigator — HammondCare; Rachael Wright, BAppSc(OccThpy), Principal Investigator — SWSLHD; Renee Fortunato, B.App.Sc.(Phys.), Principal Investigator — SWSLHD; Wei Xuan, MSc MAppStat PhD, Principal Investigator — Ingham Institute
Locations (3):
- Australia (3):
  - Braeside Hospital, Sydney, New South Wales
  - Fairfield Hospital, Sydney, New South Wales
  - Sutherland Hospital, Sydney, New South Wales

REFERENCES:
- [Derived] Buhagiar MA, Naylor JM, Harris IA, Xuan W, Kohler F, Wright R, Fortunato R. Effect of Inpatient Rehabilitation vs a Monitored Home-Based Program on Mobility in Patients With Total Knee Arthroplasty: The HIHO Randomized Clinical Trial. JAMA. 2017 Mar 14;317(10):1037-1046. doi: 10.1001/jama.2017.1224. PMID 28291891
- [Derived] Buhagiar MA, Naylor JM, Harris IA, Xuan W, Kohler F, Wright RJ, Fortunato R. Hospital Inpatient versus HOme-based rehabilitation after knee arthroplasty (The HIHO study): study protocol for a randomized controlled trial. Trials. 2013 Dec 17;14:432. doi: 10.1186/1745-6215-14-432. PMID 24341348